CLINICAL TRIAL: NCT04688931
Title: A Randomized, Controlled, Open-Label Study of the Efficacy, Durability, and Safety of UGN-102 With or Without TURBT in Patients With Low-Grade Intermediate-Risk Non-Muscle Invasive Bladder Cancer (LG-IR-NMIBC)
Brief Title: A Phase 3 Study of UGN-102 for Low-Grade Intermediate-Risk Non-Muscle Invasive Bladder Cancer
Acronym: ATLAS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Alternate approach pursued
Sponsor: UroGen Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL006
Record Dates: First submitted 2020-07-21; First posted 2020-12-30 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Bladder Cancer; Urothelial Carcinoma; Urothelial Carcinoma Bladder
Keywords: Non-muscle invasive bladder cancer; Low grade non-muscle invasive bladder cancer; Intermediate risk non-muscle invasive bladder cancer; NMIBC; UGN-102; Mitomycin; Transurethral resection of bladder tumors; TURBT
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell; Non-Muscle Invasive Bladder Neoplasms | interventions — Mitomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- UGN-102 ± TURBT (Experimental): 6 weekly intravesical instillations of UGN-102 (75 mg mitomycin) starting on Day 1 + TURBT for patients with NCR due to residual LG disease at the 3-month Visit (3 months after the start of treatment with UGN-102).
  Interventions: Drug: UGN-102; Procedure: TURBT
- TURBT Alone (Active Comparator): TURBT on Day 1 + repeat TURBT for patients with NCR due to residual LG disease at the 3-month Visit (3 months after the initial TURBT).
  Interventions: Procedure: TURBT

INTERVENTIONS:
Drug: UGN-102 — UGN-102 consists of mitomycin and sterile hydrogel (a proprietary thermally responsive gel) that is used to reconstitute mitomycin before instillation. The reverse thermal properties of UGN-102 allow for local administration of mitomycin as a liquid under chilled conditions, with subsequent conversion to a semi-solid gel depot following instillation into the bladder.
  Other Names: UGN-102 (mitomycin) for intravesical solution
  Arms: UGN-102 ± TURBT
Procedure: TURBT — The current standard of care for treatment of LG-IR-NMIBC is TURBT under general anesthesia.
  Other Names: Transurethral resection of bladder tumors

SUMMARY:
This global, randomized, controlled, open-label Phase 3 study was designed to assess the long-term efficacy and safety of UGN-102 (mitomycin) for intravesical solution with or without (±) transurethral resection of bladder tumors (TURBT) versus TURBT alone for the treatment of patients with low-grade intermediate-risk non-muscle invasive bladder cancer (LG-IR-NMIBC).

DETAILED DESCRIPTION:
Eligible patients were randomized in a 1:1 ratio to UGN-102 ± TURBT or TURBT alone. Randomization was stratified by the presence of a previous LG-NMIBC episode within 1 year of the current diagnosis (yes or no). Starting on Day 1, patients randomized to the UGN-102 ± TURBT arm will receive 6 weekly intravesical instillations of UGN-102 and patients randomized to the TURBT alone arm underwent TURBT.

All patients returned to the clinic approximately 3 months after the start of treatment for a disease assessment visit. Response to treatment was determined based on visual observation (white light cystoscopy), histopathology of any remaining or new lesions, and voiding urine cytology. Patients confirmed to have a complete response (CR), defined as having no detectable disease (NDD) in the bladder, received no further treatment and entered the Follow-up Period of the study. Patients confirmed to have a non-complete response (NCR) due to residual LG disease in either treatment arm underwent TURBT of any remaining lesions and then entered the Follow-up Period of the study.

During the Follow-up Period, patients returned to the clinic every 3 months to determine if they remained disease free. Patients remained on study until completion of all follow-up visits or until disease recurrence, disease progression, or death was documented, whichever occurred first. Patients determined to have a protocol-defined recurrence or progression at any follow-up or unscheduled visit were considered to have completed the study and released to the care of their treating physician.

Study enrollment was stopped early by the sponsor to pursue an alternative development strategy for UGN-102 in the treatment of bladder cancer. Patients who had consented at the time the trial terminated were permitted to continue, but follow-up was terminated once the last patient had been followed for 15 months after the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.
2. Patient who has newly diagnosed or historic LG-NMIBC (Ta) histologically confirmed by cold cup biopsy at Screening or within 8 weeks of Screening.
3. Has intermediate risk disease, defined as having 1 or 2 of the following:

   * Presence of multiple tumors;
   * Solitary tumor > 3 cm;
   * Recurrence (≥ 1 occurrence of LG-NMIBC within 1 year of the current diagnosis).
4. Negative voiding cytology for HG disease within 6 weeks of Screening.
5. Has adequate organ and bone marrow function as determined by the following routine laboratory tests:

   * Leukocytes ≥ 3,000 cells per μL;
   * Absolute neutrophil count ≥ 1,500 cells per μL;
   * Platelets ≥ 100,000 per μL;
   * Hemoglobin ≥ 9.0 g/dL;
   * Total bilirubin ≤ 1.5 x upper limit of normal (ULN);
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN;
   * Alkaline phosphatase (ALP) ≤ 2.5 × ULN;
   * Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min.
6. Has no evidence of active urinary tract infection (UTI).
7. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for clinical study participants. Women of childbearing potential (defined as premenopausal women who have not been sterilized), including female patients and female partners of male patients, must be willing to use 2 acceptable forms of effective contraception from enrollment through 6 months post-treatment.

Exclusion Criteria:

1. History of carcinoma in situ (CIS) on preliminary cystoscopy within 5 years of enrollment.
2. Received Bacillus Calmette-Guérin (BCG) treatment for urothelial carcinoma (UC) within previous 1 year.
3. History of HG papillary UC in the past 2 years.
4. Known allergy or sensitivity to mitomycin that in the investigator's opinion cannot be readily managed.
5. Clinically significant urethral stricture that would preclude passage of a urethral catheter.
6. History of pelvic radiotherapy.
7. History of:

   * Neurogenic bladder;
   * Active urinary retention;
   * Any other condition that would prohibit normal voiding.
8. Past or current muscle invasive (ie, T2, T3, T4) or metastatic UC or concurrent upper tract UC.
9. Current tumor stage of T1.
10. Has an underlying substance abuse or psychiatric disorder such that, in the opinion of the investigator, the patient would be unable to comply with the protocol.
11. History of prior treatment with an intravesical chemotherapeutic agent except for a single dose of chemotherapy immediately after any previous TURBT.
12. Has previously participated in a study in which they received UGN-102.
13. Has participated in a study with an investigational agent or device within 30 days of randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2021-02-19 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandip Prasad, MD, Principal Investigator — Atlantic Health System
Locations (139):
- United States (33):
  - Arizona Institute of Urology, PLLC, Tucson, Arizona
  - Loma Linda University Medical Center, Loma Linda, California
  - Urology Group of Southern California, Los Angeles, California
  - San Diego Clinical Trials, San Diego, California
  - Providence Saint John's Health Center, Santa Monica, California
  - Skyline Urology, Sherman Oaks, California
  - University of Chicago Hospital, Chicago, Illinois
  - Comprehensive Urologic Care, Lake Barrington, Illinois
  - First Urology, PSC, Jeffersonville, Indiana
  - Wichita Urology Group, Wichita, Kansas
  - Regional Urology, LLC, Shreveport, Louisiana
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Hanover, Maryland
  - Adult & Pediatric Urology, PC, Omaha, Nebraska
  - Urology Center, Las Vegas, Nevada
  - New Jersey Urology, Bloomfield, New Jersey
  - New Jersey Urology, Englewood, New Jersey
  - Garden State Urology, Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - Great Lakes Physician dba WNY Urology Associates, Cheektowaga, New York
  - AccuMed Research Associates, Garden City, New York
  - Manhattan Medical Research, New York, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Associated Medical Professionals of NY, PLLC, Syracuse, New York
  - UNC Chapel Hill Memorial Hospital, Chapel Hill, North Carolina
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Centers for Advanced Urology, LLP d.b.a Mid-Atlantic Urology, Bala-Cynwyd, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center and College of Medicine, Hershey, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Urology San Antonio, San Antonio, Texas
- Bulgaria (22):
  - Multiprofile Hospital for Active Treatment "Puls", Department of Urology, Blagoevgrad
  - Multiprofile Hospital for Active Treatment - Blagoevgrad, Blagoevgrad
  - Complex Oncology Center - Burgas, Burgas
  - Multiprofile Hospital for Active Treatment "Dr. Tota Venkova", Gabrovo, Department of Urology, Gabrovo
  - Multiprofile Hospital for Active Treatment "Sveti Nikolai Chudotvorets", Lom, Lom
  - Multiprofile Hospital for Active Treatment "City Clinic - Sveti Georgi", Montana
  - University Multiprofile Hospital for Active Treatment "Dr. Georgi Stranski", Pleven, Urology Clinic, Pleven
  - University Multiprofile Hospital for Active Treatment "Sveta Marina" - Pleven, Department of Urology, Pleven
  - Multiprofile Hospital for Active Treatment Park Hospital, Plovdiv
  - University Multiprofile Hospital for Active Treatment "Sveti Georgi", Plovdiv, Clinic of Urology, Plovdiv
  - University Multiprofile Hospital for Active Treatment, Plovdiv, Department of Urology, Plovdiv
  - University Multiprofile Hospital for Active Treatment 'Kanev', Ruse, Department of Urology, Rousse
  - Multiprofile Hospital for Active Treatment - Shumen, Shumen, Department of Urology, Shumen
  - University Multiprofile Hospital for Active Treatment "Aleksandrovska", Sofia, Urology Clinic, Sofia
  - University Multiprofile Hospital for Active Treatment and Emergency Medicine "N.I. Pirogov", Sofia, Urology Clinic, Sofia
  - Multiprofile Hospital for Active Treatment - Targovishte, Targovishte
  - Multiprofile Hospital for Active Treatment, Varna part of Military Medical Academy, Clinic of Urology, Varna
  - Multiprofile Hospital for Active Treatment "Sveta Anna", Varna, Urology Clinic, Varna
  - University Multiprofile Hospital for Active Treatment "Sveta Marina", Varna
  - Multiprofile Regional Hospital for Active Treatment "Dr. Stefan Cherkezov", Veliko Tarnovo, Department of Urology, Veliko Tarnovo
  - First Private Hospital Vratsa, Department of Urology, Vratsa
  - Multiprofile Hospital for Active Treatment "Sveti Pantaleymon", Yambol, Department of Urology, Yambol
- Estonia (5):
  - East Viru Central Hospital, Surgery Clinic, Kohtla-Järve
  - East Tallinn Central Hospital Ltd., Surgery Clinic, Centre of Urology, Tallinn
  - West Tallinn Central Hospital Ltd., Department of Urology, Tallinn
  - North Estonia Medical Centre Foundation Ltd., Surgery Clinic, General and Oncology Urology Centre, Tallinn
  - Tartu University Hospital, Surgery Clinic, Department of Urology and Kidney Transplantation, Tartu
- Georgia (9):
  - LTD Central University Clinic After Academic N. Kipshidze, Tbilisi
  - JSC Jerarsi, Department of Urology, Tbilisi
  - LTD Acad. F. Todua Medical Center - LTD Research Institute of Clinical Medicine, Clinical Research Department, Tbilisi
  - LTD Gidmedi, Urology Department, Tbilisi
  - LTD L. Managadze National Center of Urology, Department of Urology, Tbilisi
  - LTD MMT Hospital, Urology Department, Tbilisi
  - Malkhaz Katsiashvili Multiprofile Emergency Medicine Center LTD, Department of Urology, Tbilisi
  - Pineo Medical Ecosystem Ltd., Department of Urology, Tbilisi
  - Tbilisi State Medical University and Ingorokva High Technology Medical Center University Clinic LTD, Urology Department, Tbilisi
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Latvia (4):
  - Liepajas Regional Hospital, Urology Department, Liepāja
  - P. Stradins Clinical University Hospital, Center for Urology, Riga
  - LLC Riga East University Hospital, Clinic of Urology and Oncologic Urology, Riga
  - Daugavpils Regional Hospital, Urology Department, Riga
- Poland (6):
  - Jan Biziel University Hospital #2 in Bydgoszcz, Teaching Department of Urology, Bydgoszcz
  - AKMED, Gliwice
  - Prof.E Michalowski Specialist Hospital, Katowice
  - SCM sp. z o.o. (LLC), Krakow
  - "City Clinic" Limited Liability Company, Warsaw
  - Miedzyleski Specialist Hospital in Warsaw, Department of Urology, Warsaw
- Russia (27):
  - Krasnoyarsk A.I. Kryzhanovsky Regional Oncology Center, Krasnoyarsk
  - D.D. Pletnyov City Clinical Hospital, Department of Oncourology, Moscow
  - Moscow City Oncology Hospital #62, Moscow
  - Murmansk Bayandin Regional Clinical Hospital, Murmansk
  - Privolzhsky Regional Medical Center, Urology Department, Nizhny Novgorod
  - Tsyb Medical Radiology Research Center, Oncourology Department, Obninsk
  - Clinical Oncology Center, Department of Urology and Oncology, Omsk
  - N.N. Burdenko Penza Regional Clinical Hospital, Department of Urology, Penza
  - Pyatigorsk City Clinical Hospital, Department of Urology, Pyatigorsk
  - Leningrad Regional Clinical Oncology Center, Department of Chemotherapy, Saint Petersburg
  - Aleksandrovskaya City Hospital, Department of Urology, Saint Petersburg
  - St. Petersburg Clinical Hospital under the Russian Academy of Sciences, Department of Urology, Saint Petersburg
  - A.M. Nikiforov Russian Center for Emergency and Radiology Medicine, Department of Urology, Saint Petersburg
  - St. Luka Clinical Hospital, Department of Urology, Saint Petersburg
  - St.-Petersburg Scientific Research Institute of Phthisiopulmonology, Saint Petersburg
  - Medical and Sanitary Unit #70 of "Passazhiravtotrans", Saint Petersburg
  - I.I. Mechnikov North-Western State Medical University, Department of Urology, Saint Petersburg
  - Railway Clinical Hospital under OAO Russian Railways, Saint Petersburg
  - First I.P. Pavlov State Medical University of St. Petersburg, Saint Petersburg
  - N.N. Petrov National Medical Research Center of Oncology, Oncourology Department, Saint Petersburg
  - City Hospital #15, Urology Department #12, Saint Petersburg
  - Siberian State Medical University, Tomsk
  - Regional Oncology Center, Tyumen, Oncology Department, Tyumen
  - Republican Clinical Oncology Center, Ufa
  - Volgograd Regional Center for Urology and Nephrology, Urology Department, Volzhskiy
  - Medical Center for Diagnostics and Prevention Plus, Yaroslavl
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg
- Serbia (4):
  - Clinical Center of Serbia, Clinic of Urology, Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Clinic of Surgery, Department of Urology, Belgrade
  - Clinical Hospital Center Zemun, Urology unit, Belgrade
  - Clinical Center Kragujevac, Clinic of Urology, Nephrology and Dialysis, Kragujevac
- Ukraine (24):
  - Chernihiv Medical Center of Modern Oncology, Chernihiv
  - Regional Communal Noncommercial Enterprise: Chernivtsi Regional Clinical Hospital, Chernivtsi
  - Regional Municipal Non-commercial Enterprise "Chernivtsi Emergency Medical Hospital", Urology Department, Chernivtsi
  - Public Enterprise "Dnipropetrovsk I.I. Mechnikov Regional Clinical Hospital" under Dnipropetrovsk Regional Council, Urology Department #2, Dnipro
  - Public Non-Profit Enterprise "City Clinical Hospital #6" under Dnipro City Council, Department of Urology, Dnipro
  - Public Non-Profit Enterprise "City Clinical Hospital #4" under Dnipro City Council, Department of Geriatric Urology Care, Dnipro
  - Public Non-Profit Enterprise "Regional Clinical Hospital under Ivano-Frankivsk Regional Council", Department of Urology, Ivano-Frankivsk
  - Prykarpattia Clinical Oncology Center under Ivano-Frankivsk Regional Council, Ivano-Frankivsk
  - Public Non-Profit Enterprise under Kharkiv Regional Council "V.I. Shapoval Regional Medical Clinical Center for Urology and Nephrology", Urology Department #5, Kharkiv
  - Communal Non-Profit Enterprise "Regional Center of Oncology", Department of Oncourology, Kharkiv
  - Public Non-Profit Enterprise under Kharkiv Regional Council "Regional Clinical Specialized Center for Radiation Protection of Population", Department of Surgery, Kharkiv
  - Communal non-commercial enterprise of Kherson regional council "Kherson regional oncological dispensary", Kherson
  - State Institution: Institute of Urology under the National Academy of Medical Sciences of Ukraine, Kyiv
  - Volyn Regional Medical Oncology Centre, Lutsk
  - Communal Noncommercial Enterprise of Lviv Regional Council "Lviv Regional Clinical Hospital", Department of Urology, Lviv
  - Public Non-profit Enterprise under Lviv Regional Council: Lviv Regional Treatment and Diagnostics Oncology Center, Lviv
  - Municipal Non-Profit Enterprise "Lviv Clinical Emergency Care Hospital", Department of Urology, Lviv
  - Public Non-Profit Enterprise "Odesa Regional Clinical Hospital" under Odesa Regional Council, Odesa
  - Public Non-Profit Enterprise "City Clinical Hospital #10" under Odesa City Council, Department of Urology and Nephrology, Odesa
  - Sumy Regional Clinical Oncology Center, Sumy
  - Public Non-Profit Enterprise Ternopil Regional Clinical Oncology Center, Department of Chemotherapy, Ternopil
  - Municipal non-profit enterprise "Transcarpathian antitumor center" of the Transcarpathian Regional Council, Uzhhorod
  - Communal Nonprofit Enterprise "Podilsky Regional Center of Oncology of Vinnytsia Regional Council", Vinnytsia
  - Municipal Nonprofit Enterprise: Zaporizhia Regional Clinical Hospital under Zaporizhia Regional Council, Department of Urology, Zaporizhia

REFERENCES:
- [Result] Prasad SM, Huang WC, Shore ND, Hu B, Bjurlin M, Brown G, Genov P, Shishkov D, Khuskivadze A, Ganev T, Marchev D, Orlov I, Kopyltsov E, Zubarev V, Nosov A, Komlev D, Burger B, Raju S, Meads A, Schoenberg M. Treatment of Low-grade Intermediate-risk Nonmuscle-invasive Bladder Cancer With UGN-102 +/- Transurethral Resection of Bladder Tumor Compared to Transurethral Resection of Bladder Tumor Monotherapy: A Randomized, Controlled, Phase 3 Trial (ATLAS). J Urol. 2023 Oct;210(4):619-629. doi: 10.1097/JU.0000000000003645. Epub 2023 Aug 7. PMID 37548555

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | UGN-102 ± TURBT | TURBT Alone
Started | 142 | 140
Completed | 123 | 106
Not Completed | 19 | 34
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 5 | 16
Not completed — Physician Decision | 3 | 5
Not completed — Noncompliance | 0 | 1
Not completed — Lost to Follow-up | 1 | 3
Not completed — Randomization Error | 3 | 0
Not completed — Not Eligible | 1 | 3
Not completed — Disease Progression | 0 | 2
Not completed — Sponsor Requirement | 1 | 1
Not completed — Other Reason | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UGN-102 ± TURBT | TURBT Alone | Total
Number analyzed (Participants) | 142 | 140 | 282
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 63 | 114
  >=65 years | 91 | 77 | 168
Age, Continuous [Median (Full Range); unit: years] | 68 [23 to 85] | 67 [29 to 88] | 68 [23 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 47 | 84
  Male | 105 | 93 | 198
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 140 | 137 | 277
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 140 | 139 | 279
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Latvia | 9 | 7 | 16
  United States | 14 | 11 | 25
  Ukraine | 11 | 20 | 31
  Poland | 1 | 1 | 2
  Georgia | 15 | 15 | 30
  Israel | 0 | 1 | 1
  Bulgaria | 37 | 26 | 63
  Serbia | 1 | 4 | 5
  Estonia | 10 | 8 | 18
  Russia | 44 | 47 | 91
Previous LG-NMIBC Episode(s) [Count of Participants; unit: Participants]
  Yes | 54 | 65 | 119
  No | 88 | 75 | 163
Previous LG-NMIBC Episode(s) Within 1 Year [Count of Participants; unit: Participants]
  Yes | 41 | 40 | 81
  No | 101 | 100 | 201
Prior TURBT(s) [Count of Participants; unit: Participants]
  Yes | 52 | 64 | 116
  No | 90 | 76 | 166
Tumor Size [Count of Participants; unit: Participants]
  ≤ 3 cm | 69 | 73 | 142
  > 3 cm | 67 | 59 | 126
  Missing | 6 | 8 | 14
Tumor Count [Count of Participants; unit: Participants]
  Multiple | 82 | 94 | 176
  Single | 54 | 40 | 94
  Missing | 6 | 6 | 12
Smoking History [Count of Participants; unit: Participants]
  Non-smoker | 63 | 73 | 136
  Smoker | 79 | 67 | 146

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS)
Description: DFS is defined as the time from randomization until the earliest date of any of the following events: failure to be rendered free of local disease at the 3-month Visit (TURBT arm only), recurrence of LG disease after the 3-month Visit (ie, during the Follow-up Period), progression to high-grade (HG) disease, or death due to any cause. Summarized is the Kaplan-Meier estimated probability of remaining event-free at 15 months from randomization.
Time Frame: 15 months
Population: All randomized patients regardless of whether the treatment was administered.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UGN-102 ± TURBT | TURBT Alone
Number analyzed (Participants) | 142 | 140
percentage of participants | 72.0 [63.1 to 79.2] | 49.5 [39.6 to 58.6]
Statistical Analysis 1: Comparison: UGN-102 ± TURBT vs TURBT Alone; Test type: Other — The analysis is descriptive in nature; Cox Proportional Hazard = 0.45, 95% CI 2-sided [0.29 to 0.68] — The hazard ratio represents the relative risk of having an event in the treatment arm (numerator) versus the control arm (denominator)

2. Secondary Outcome: Time to Recurrence (TTR)
Description: TTR is defined as the time from randomization until the earliest date of any of the following events: failure to be rendered free of local disease at the 3-month Visit (TURBT arm only), recurrence of LG disease after the 3-month Visit (ie, during the Follow-up Period), or progression to HG disease. Summarized is the Kaplan-Meier estimated probability of remaining event-free at 15 months from randomization.
Time Frame: 15 months
Population: All randomized patients regardless of whether the treatment was administered.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UGN-102 ± TURBT | TURBT Alone
Number analyzed (Participants) | 142 | 140
percentage of participants | 72.0 [63.1 to 79.2] | 50.3 [40.4 to 59.4]
Statistical Analysis 1: Comparison: UGN-102 ± TURBT vs TURBT Alone; Test type: Other — The analysis is descriptive in nature; Cox Proportional Hazard = 0.46, 95% CI 2-sided [0.30 to 0.70] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Complete Response Rate (CRR)
Description: CRR is defined as the percentage of patients who achieve CR at the 3-month Visit.
Time Frame: 3 months
Population: All randomized patients regardless of whether the treatment was administered. At the time of the 3-month Visit, patients had received only the primary intervention (6 weekly intravesical instillations of UGN-102 starting on Day 1 or TURBT on Day 1).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- UGN-102: 6 weekly intravesical instillations of UGN-102 (75 mg mitomycin) starting on Day 1.
- TURBT Alone: TURBT on Day 1.
Arm/Group | UGN-102 | TURBT Alone
Number analyzed (Participants) | 142 | 140
percentage of participants | 64.8 [56.3 to 72.6] | 63.6 [55.0 to 71.5]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from first documented CR until the earliest date of recurrence of LG disease, progression to HG disease, or death due to any cause. DOR applies only to patients who achieve CR at the 3-month Visit. Summarized is the Kaplan-Meier estimated probability of remaining in response at 12 months after 3-month CR.
Time Frame: 12 months
Population: All patients who achieved CR at the 3-month disease assessment. Patients who achieved CR at 3 months received only the primary intervention (6 weekly intravesical instillations of UGN-102 starting on Day 1 or TURBT on Day 1).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UGN-102 | TURBT Alone
Number analyzed (Participants) | 92 | 89
percentage of participants | 79.7 [69.3 to 86.9] | 67.7 [55.8 to 77.1]
Statistical Analysis 1: Comparison: UGN-102 vs TURBT Alone; Test type: Other — The analysis is descriptive in nature; Cox Proportional Hazard = 0.46, 95% CI 2-sided [0.24 to 0.86] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Observed CRR at Scheduled Disease Assessment Time Points
Description: Observed CRR at scheduled disease assessment time points is defined as the percentage of patients who achieve CR at the 3-month Visit and maintain CR up to a particular follow-up visit. Summarized is the observed percentage of patients remaining in response at 3, 6, 9, and 12 months after 3-month CR.
Time Frame: 12 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | UGN-102 | TURBT Alone
Number analyzed (Participants) | 92 | 89
percentage of participants
  3 Months After 3-Month CR | 92.4 [84.9 to 96.9] | 71.9 [61.4 to 80.9]
  6 Months After 3-Month CR | 80.4 [70.9 to 88.0] | 62.9 [52.0 to 72.9]
  9 Months After 3-Month CR | 75.0 [64.9 to 83.4] | 57.3 [46.4 to 67.7]
  12 Months After 3-Month CR | 71.7 [61.4 to 80.6] | 55.1 [44.1 to 65.6]

6. Secondary Outcome: Number of TURBTs
Description: Number of TURBTs is defined as the average number of per protocol TURBTs per patient in each arm. Per protocol TURBTs are defined as the Day 1 TURBT for patients in the TURBT alone arm and TURBT due to residual LG disease at the 3-month disease assessment in either arm.
Time Frame: 3 months
Population: All patients who received any dose of UGN-102 (treatment arm) or at least one TURBT intervention (control arm).
Measure: Mean (Standard Deviation); unit: TURBT procedures
Arm/Group | UGN-102 ± TURBT | TURBT Alone
Number analyzed (Participants) | 138 | 132
TURBT procedures | 0.2 (0.38) | 1.1 (0.34)

7. Secondary Outcome: Changes From Baseline in Health-related Quality of Life
Description: The European Organisation for Research and Treatment of Cancer (EORTC) 24-item quality of life questionnaire for patients with NMIBC (QLQ-NMIBC24) is a patient-reported instrument that assesses 11 domains (urinary symptoms, malaise, future worries, bloating and flatulence, intravesical treatment issues, sexual intimacy, risk of contaminating partner, male sexual problems, female sexual problems, sexual function, and sexual enjoyment).
  All of the domains range in score from 0 to 100 with lower scores reflecting better functioning/quality of life and higher scores reflecting worse functioning/quality of life.
  Summarized is the change from baseline in domain scores at the 3-month Visit. Changes in domain scores were calculated for patients with non-missing answers at both time points.
Time Frame: Pre-treatment to 3 months after the start of treatment
Population: All patients who received any dose of UGN-102 (treatment arm) or at least one TURBT intervention (control arm). At the time of the 3-month Visit, patients had received only the primary intervention (6 weekly intravesical instillations of UGN-102 starting on Day 1 or TURBT on Day 1).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UGN-102 | TURBT Alone
Number analyzed (Participants) | 138 | 132
score on a scale
  Urinary Symptoms: number analyzed (Participants) | 125 | 116
  Urinary Symptoms | -10.7 (17.88) | -4.5 (20.04)
  Malaise: number analyzed (Participants) | 125 | 116
  Malaise | -4.4 (13.58) | -1.1 (16.41)
  Intravesical Treatment Issues: number analyzed (Participants) | 125 | 116
  Intravesical Treatment Issues | -4.0 (25.61) | -2.9 (25.09)
  Future Worries: number analyzed (Participants) | 125 | 116
  Future Worries | -12.7 (26.49) | -8.3 (26.74)
  Bloating and Flatulence: number analyzed (Participants) | 125 | 116
  Bloating and Flatulence | -7.7 (18.03) | -3.0 (16.68)
  Male Sexual Problems: number analyzed (Participants) | 91 | 80
  Male Sexual Problems | 0.9 (32.99) | -0.6 (30.75)
  Sexual Intimacy: number analyzed (Participants) | 63 | 65
  Sexual Intimacy | 0.0 (19.86) | 3.6 (30.12)
  Risk of Contaminating Partner: number analyzed (Participants) | 61 | 64
  Risk of Contaminating Partner | 1.6 (26.12) | 0.0 (16.80)
  Female Sexual Problems: number analyzed (Participants) | 10 | 15
  Female Sexual Problems | -10.0 (16.10) | -8.9 (15.26)
  Sexual Function: number analyzed (Participants) | 125 | 116
  Sexual Function | 0.4 (18.02) | -1.6 (22.20)
  Sexual Enjoyment: number analyzed (Participants) | 61 | 65
  Sexual Enjoyment | 8.7 (36.97) | -1.0 (32.26)

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, and TEAEs of Special Interest
Description: The number of patients with each type of event will be summarized. TEAEs were defined as adverse events (AEs) that occurred on or after the day of first instillation of UGN-102 for patients in the UGN-102 ± TURBT arm or the day of initial TURBT for patients in the TURBT alone arm, or pre-treatment events that worsened during the study.
Time Frame: Up to 21 months
Population: All patients who received any dose of UGN-102 (treatment arm) or at least one TURBT intervention (control arm).
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102 ± TURBT | TURBT Alone
Number analyzed (Participants) | 138 | 132
Participants
  Any TEAEs | 104 | 63
  Any serious TEAEs | 12 | 7
  Any TEAEs of special interest | 78 | 36

9. Secondary Outcome: Number of Participants With Post-baseline Potentially Clinically Significant (PCS) Hematology Values
Description: The number of patients with each type of event will be summarized.
Time Frame: Up to 6 months
Population: All patients who received any dose of UGN-102 (treatment arm) or at least one TURBT intervention (control arm) and who had non-missing laboratory values at the specified time.
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102 ± TURBT | TURBT Alone
Number analyzed (Participants) | 138 | 126
Participants
  Hemoglobin < 0.8 × lower limit of normal and > 20% decrease from baseline | 4 | 1
  Leukocytes ≤ 2.8 × 10^3/μL | 4 | 1
  Leukocytes ≥ 16.0 × 10^3/μL | 1 | 0
  Platelets < 75 × 10^3/μL | 1 | 0

10. Secondary Outcome: Number of Participants With Post-baseline PCS Serum Chemistry Values
Description: The number of patients with each type of event will be summarized.
Time Frame: Up to 6 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | UGN-102 ± TURBT | TURBT Alone
Number analyzed (Participants) | 138 | 126
Participants
  Alanine aminotransferase > 3 × upper limit of normal (ULN) | 2 | 1
  Aspartate aminotransferase > 3 × ULN | 2 | 1
  Bilirubin > 1.5 × ULN | 3 | 2
  Creatinine > 2.2 mg/dL | 0 | 1
  Gamma glutamyl transferase > 2.5 × ULN | 5 | 1
  Potassium < 3.0 mEq/L | 0 | 1
  Potassium > 5.5 mEq/L | 18 | 10
  Sodium ≤ 130 mEq/L | 2 | 1
  Sodium > 150 mEq/L | 2 | 0

ADVERSE EVENTS:
Time Frame: Up to 21 months
Description: Per protocol, sites were instructed to report AEs that occurred from the signing of the informed consent form to the 6-month Visit. After the 6-month Visit, all serious AEs (regardless of causality) and non-serious AEs assessed as related to study treatment (UGN-102 or TURBT) or study procedures were to be reported until the End of Study Visit.
Arm/Group | UGN-102 ± TURBT | TURBT Alone
All-Cause Mortality (participants affected / at risk) | 0/138 | 1/132
Serious Adverse Events (participants affected / at risk) | 12/138 | 7/132
Other Adverse Events (participants affected / at risk) | 102/138 | 62/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UGN-102 ± TURBT (N=138) | TURBT Alone (N=132)
COVID-19 (Infections and infestations) | 4 | 2
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 2
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UGN-102 ± TURBT (N=138) | TURBT Alone (N=132)
Dysuria (Renal and urinary disorders) | 42 | 6
Micturition urgency (Renal and urinary disorders) | 25 | 10
Nocturia (Renal and urinary disorders) | 25 | 9
Pollakiuria (Renal and urinary disorders) | 22 | 8
Haematuria (Renal and urinary disorders) | 9 | 5
Flatulence (Gastrointestinal disorders) | 13 | 4
Abdominal distension (Gastrointestinal disorders) | 6 | 4
COVID-19 (Infections and infestations) | 7 | 6
Cystitis (Infections and infestations) | 5 | 5
Urinary tract infection (Infections and infestations) | 4 | 5
Malaise (General disorders) | 8 | 2
Fatigue (General disorders) | 5 | 0
Pyrexia (General disorders) | 5 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 9 | 4
Headache (Nervous system disorders) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT04688931/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT04688931/SAP_001.pdf